CLINICAL TRIAL: NCT03326115
Title: Effectiveness of a Peer Visitation Program to Improve Patient Activation and Functional Outcomes and Quality of Life During Amputation Rehabilitation
Brief Title: Effectiveness of a Peer Visitation Program to Improve Patient Activation and Quality of Life During Amputation Rehabilitation
Acronym: AC PVP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prosthetic Design & Research (Industry)
Collaborators: Amputee Coalition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AC PVP
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Amputation
Keywords: patient activation; peer visitation; amputee
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Visitation Program (PVP) (Experimental): Participants in this group will begin participation in the Peer Visitation Program (PVP) beginning at amputation date with the initiation window ranging from immediately pre-operative to 7 days post operative.
  Interventions: Behavioral: Peer Visitation Program
- Delayed Peer Visitation (NoPVP) (No Intervention): Not participating in a Peer Visitation Program for 60 days post-operatively, followed by participation and completion in a PVP 60 days later than the PVP group for a total of 120 days.

INTERVENTIONS:
Behavioral: Peer Visitation Program — The Amputee Coalition's Peer Visitation Program (PVP) trains amputee peer supporters to properly navigate a new or less-experienced amputee through the process of rehabilitation. Peer support plays an important role, following the amputation of a limb, by allowing patients to meet other amputees and discuss lifestyle changes post-amputation. Subjects randomized to the PVP group will receive the intervention (visitation by a Certified Peer Visitor) immediately at amputation. Subjects randomized to the non-PVP group will not receive CPV visits immediately at amputation. Rather, they will receive delayed PVP intervention beginning 60 days after amputation and lasting a total of 60 days (or at 120 days post-amputation).
  Arms: Peer Visitation Program (PVP)

SUMMARY:
There is no known interventional clinical trial evidence for existing support and the reintegration strategy of a peer visitation program following amputation. The Amputee Coalition Peer Visitation Program is the only national and VA recognized program for amputees, however, it has not been rigorously tested for effectiveness. Therefore, the objective of this study is to demonstrate the Amputee Coalition Peer Visitation Program (AC PVP) will improve functional outcomes for Service Members, Veterans, and civilians during amputation rehabilitation.

DETAILED DESCRIPTION:
In the fields of medicine and public health management, navigation and peer visitation programs consider patients as are their own important resources, who should be actively involved in the health care organization and throughout the process of care delivery and rehabilitation. The importance of promoting a more active role of patients in the management of their own health care is recognized by health care experts, managers, and policy makers. Programs that engage patients in their own health care are reported as an important strategy to improve adherence, outcomes, satisfaction toward the health care provider, and reduction of health care costs. The emotional adjustment to an amputation is sometimes the most challenging part. Peer visitation allows the patient to speak directly with another amputee who has shared a similar experience, allowing them to relate feelings and concerns about the loss of a limb to someone who has already endured the process and lives with the condition daily.

There is increasing national and international interest in patient education programs. The ultimate anticipated outcome for individuals attending these programs is improvement in quality of life. Patient empowerment, self-efficacy, and self-management have also been found to be key intermediate outcomes of acute amputation rehabilitation, but have been somewhat difficult to operationalize, measure, and subsequently report in terms of patient impact. There is no known interventional clinical trial evidence for existing support and the reintegration strategy of a peer visitation program following amputation.

The Amputee Coalition Peer Visitation Program is the only national and VA recognized program for amputees, however, it has not been rigorously tested for effectiveness. Therefore, the objective of this study is to demonstrate the Amputee Coalition Peer Visitation Program (AC PVP) will improve functional outcomes for Service Members, Veterans, and civilians during amputation rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Any candidate for lower extremity amputation
* Any immediate post operative lower extremity amputation within 7 days of amputation
* Willing and able to comply with the study protocol
* Able to provide informed consent
* Male or female, of any ethnicity
* 18 - 75 years of age
* Any body weight

Exclusion Criteria:

* Any level of amputation other than lower extremity
* Known cognitive impairment
* Does not speak English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Function/Quality of Life - PVP Group | 60 days post-amputation
  The MOS short-form health survey (SF-36) will be used to measure function. The SF-36 measures health status in eight dimensions: physical functioning; role limitations due to physical health problems; bodily pain; general health perceptions; vitality, energy, and fatigue; social functioning; role limitations due to emotional problems; and general mental health covering psychological distress and well-being. Scoring instructions from RAND Health provide guidance regarding scoring for each item in the survey and which items measure the aforementioned items.
Function/Quality of Life -NoPVP group | 120 days post-amputation
  The MOS short-form health survey (SF-36) will be used to measure function.The SF-36 measures health status in eight dimensions: physical functioning; role limitations due to physical health problems; bodily pain; general health perceptions; vitality, energy, and fatigue; social functioning; role limitations due to emotional problems; and general mental health covering psychological distress and well-being. Scoring instructions from RAND Health provide guidance regarding scoring for each item in the survey and which items measure the aforementioned items.
Depression - PVP group | 60 days post-amputation
  Depression is a treatable disorder associated commonly with amputation and can impact function and quality of life. The Patient Health Questionnaire (PHQ-9) is a questionnaire that can be entirely self-administered by the patient and interpreted by clinicians. The PHQ, a freely available instrument, assesses 8 diagnoses divided into threshold disorders and sub-threshold disorders
Depression - NoPVP group | 120 days post-amputation
  Depression is a treatable disorder associated commonly with amputation and can impact function and quality of life. The Patient Health Questionnaire (PHQ-9) is a questionnaire that can be entirely self-administered by the patient and interpreted by clinicians. The PHQ, a freely available instrument, assesses 8 diagnoses divided into threshold disorders and sub-threshold disorders
Patient Activation - PVP Group | 60 days post-amputation
  Patient activation will be measured using the Patient Activation Measure (PAM), which is an outcome measure with strong psychometric properties in chronic illness and is able to detect the level of patient activation towards their care management
Patient Activation - NoPVP Group | 120 days post-amputation
  Patient activation will be measured using the Patient Activation Measure (PAM), which is an outcome measure with strong psychometric properties in chronic illness and is able to detect the level of patient activation towards their care management

IPD SHARING:
Plan to Share IPD: No